CLINICAL TRIAL: NCT06459271
Title: A Feasibility Trial of Managing Cancer and Living Meaningfully (CALM) in Patients With Newly Diagnosed and Recurrent Advanced Ovarian Cancer
Brief Title: Feasibility of CALM in Patients With Ovarian Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-5885
Record Dates: First submitted 2024-06-05; First posted 2024-06-14 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Patient Satisfaction; Ovarian Cancer
Keywords: ovarian cancer; psychological care; CALM; psychotherapeutic intervention; psychological distress
MeSH Terms: conditions — Patient Satisfaction; Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: All participants (patients with newly diagnosed and recently recurred ovarian cancer) will receive the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Newly Diagnosed + Recently Recurred (Experimental): n = 50 patients with ovarian cancer (stage III or IV) will be enrolled in the study (25 newly diagnosed and 25 recently recurred).
  Interventions: Other: Managing Cancer And Living Meaningfully (CALM)

INTERVENTIONS:
Other: Managing Cancer And Living Meaningfully (CALM) — Our team has developed a brief, manualized, individual and couple-based psychotherapeutic intervention for patients living with advanced cancer and their primary caregivers called Managing Cancer and Living Meaningfully (CALM). CALM is a brief supportive-expressive therapy consisting of 3-6 sessions of 30-60 minutes delivered over the course of 3-6 months. This tailored therapy is focused on the most common challenges and concerns facing individuals living with advanced cancer. These four broad content domains are: 1) symptom management and communication with healthcare providers; 2) changes in self and in relationships with close others; 3) sense of meaning and purpose in life; and 4) hopes and fears about the future and mortality. The aim is to offer patients and caregivers reflective space and a supportive environment to reflect on and process the various practical and profound aspects of their life while facing advanced illness.

SUMMARY:
The goal of this feasibility trial is to determine the feasibility and acceptability of implementing a brief evidence-based psychotherapeutic intervention, Managing Cancer And Living Meaningfully (CALM), at the time of a new diagnosis and recurrence of ovarian cancer (OC).

The main questions are:

1. Is it feasible and acceptable to implement CALM for patients with newly diagnosed or recently recurred advanced OC
2. What are the prevalence and correlates of traumatic stress symptoms at baseline in patients with newly diagnosed or recently recurred advanced OC

Participants will be asked to complete questionnaires at baseline and at 3 and 6 months following a diagnosis or recurrence of stage III or IV OC. Participants will also be invited to participate in 3-6 sessions of CALM therapy.

DETAILED DESCRIPTION:
While CALM has demonstrated effectiveness in reducing depression, death anxiety and increasing preparation for end of life among patients with advanced cancer later in the illness trajectory, its feasibility and effectiveness in addressing traumatic stress symptoms (TSS) soon after a diagnosis of advanced cancer has not previously been established. Findings of this study could inform the potential development of a larger randomized effectiveness trial. This study will involve a multi-method, single-arm, feasibility trial, approaching a total of 100 OC patients (50 newly diagnosed and 50 recently recurred) at Princess Margaret Cancer Centre (PM). Measurements will be administered at baseline, 3 months and 6 months. Participants who declined to participate in the intervention will be invited to share their reasons for opting out, contributing valuable insights to our records. A subset of purposefully sampled participants will also complete qualitative interviews following the completion of outcome measures at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* new diagnosis or recurrence of stage III or stage IV OC;
* age ≥18 years
* able to complete outcome measures and engage in CALM in English.

Exclusion Criteria:

* evidence of cognitive impairment indicated in the medical record, communicated by the OC clinic team, or determined by research staff at recruitment;
* receiving psychological or psychiatric counseling from the Department of Supportive Care at PM at the time of recruitment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
Stanford Acute Stress Reaction Questionnaire (SASRQ) | This questionnaire will be administered at all timepoints (baseline, 3 months and 6 months)
  The SASRQ is a self-reported DSM-IV correspondent scale to measure a range of symptoms associated with Acute Stress Disorder (ASD), encompassing dissociation, trauma re-experiencing, avoidance behaviours, anxiety, hyperarousal, and functional impairment. The SASRQ consists of 30-items utilizing a 6-point scale that ranges from 0=not experienced to 4=very often experienced. Demonstrating robust psychometric properties, including strong test-retest reliability and consistent evidence of predictive, construct, discriminant, and convergent validity across varied populations, the SASRQ serves as a reliable and valid tool for assessment.
Clinical Evaluation Questionnaire (CEQ)-CALM | This questionnaire will be administered at 3 months and 6 months only.
  The CEQ is a 7-item validated questionnaire, created by our research team to assess the perceived benefit of interactions with health care providers in domains relevant to advanced cancer.

SECONDARY OUTCOMES:
Modified Experiences in Close Relationships (ECR-M-16) | This questionnaire will be administered at baseline.
  The ECR-M-16 is a validated measure with 16-items, has been thoughtfully adapted to be less time-consuming and alleviate any potential burden for patients who may be physically unwell.
Condensed Memorial Symptom Assessment Scale (CMSAS) | This questionnaire will be administered at all timepoints (baseline, 3 months and 6 months).
  The CMSAS CMSAS stands as a straightforward and validated self-report evaluation tool, comprising 14 items. It effectively gauges various aspects such as energy level, dry mouth, appetite, weight loss, pain, nausea, drowsiness etc. These facets are organized into three subscales: physical, psychological and symptom distress.
Patient Health Questionnaire (PHQ-9) | This questionnaire will be administered at all timepoints (baseline, 3 months and 6 months).
  The PHQ-9 is a diagnostic tool used in primary care settings to establish criteria-based diagnoses for depression. PHQ-9 is a 9-tem, self-reported questionnaire which consists of the 9 depression criteria which is highlighted within the DSM-IV. PHQ-9 is particularly favoured due to its concise structure, which efficiently identifies the presence of depressive disorders and is also able to rate the severity of depressive symptoms.
Death and Dying Distress Scale (DADDS) | This questionnaire will be administered at all timepoints (baseline, 3 months and 6 months).
  The DADDS is a tool used to evaluate the distress caused by a patients thoughts on death and dying over the previous two weeks. DADDS is a 15-items questionnaire with the aims of alleviating the fear of death and fostering psychological development (Nissim et al., 2011; Shapiro et al., 2021).The validity of DADDS has been rigorously established, with factor analysis demonstrating distress related to two factors: Finitude and Dying.

CONTACTS AND LOCATIONS:
Overall Officials: Gary M Rodin, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT06459271/Prot_SAP_000.pdf